CLINICAL TRIAL: NCT04774666
Title: Caregiver-Assisted Oral Fluid-based HIV Screening in Children: Estimation of Acceptability, Feasibility and Effectiveness Linked to Index Testing Services in Uganda
Brief Title: Caregiver-Assisted Oral Fluid-based HIV Screening in Children: Uganda
Status: Completed | Type: Observational
Sponsor: Catholic Relief Services (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CDC IRB 7292
Record Dates: First submitted 2021-02-09; First posted 2021-03-01 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: HIV Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Acceptability of OraQuick Advance© Rapid HIV-1/2 Antibody screening — Oral fluid-based HIV test

SUMMARY:
The purpose of this study is to evaluate the acceptability, feasibility and effectiveness of a caregiver-assisted oral fluid-based HIV test to screen children for HIV. The results of this study are intended to support expanded access to HIV testing and treatment services for children, and to ensure that all newly diagnosed children are linked to clinical care.

DETAILED DESCRIPTION:
Rationale: Globally, there are 1.8 million children living with HIV (CLHIV), however, despite great progress over the past 15 years, only 52% are receiving antiretroviral therapy (ART), leaving approximately 864,000 children in need of treatment.1 Pediatric case finding is the first, critical step to close the pediatric ART gap. In Uganda, there are an estimated 36,873 CLHIV in need of HIV treatment.2 Reaching this population is challenging, because children are dependent on parents and caregivers to access HIV testing services. Parents and caregivers often face logistical, societal and other barriers that limit the uptake of testing services for children. In order to achieve the second and third UNAIDS 95 targets for pediatric HIV treatment coverage and viral load suppression to reach epidemic control, country programs need to utilize increasingly targeted and innovative testing modalities to optimize the identification CLHIV. Oral fluid-based screening may present a safe, convenient and reliable way to identify CLHIV that can expand access to essential testing services in resource-limited settings where most CLHIV reside.

Methods: The study will use a cross-sectional cluster sampling design, in which 32 facilities in 16 districts will be selected using probability-proportional-to-size (PPS) sampling. In the 32 selected facilities, index parent/caregivers of approximately 4,687 children will be recruited to accept test kits for their children. Adult index parent/caregivers will be consented to participate in the study and asked for parental permission for their child(ren) to participate, given a number of oral screening kits corresponding to the number of children eligible for screening, and followed-up to confirm the oral fluid-based screening results and participate in a testing experience survey. Any children who screen HIV reactive will receive confirmatory testing and active linkage to care and treatment services. A cost analysis which includes savings associated with facility or home-based costs averted, using existing sources to estimate the costs of facility-based testing and home-based by a community health worker (CHW), preferably from antenatal settings will be undertaken.

ELIGIBILITY:
Inclusion Criteria for Index parent/caregivers:

* HIV-positive diagnosis
* 18 years old or older
* Emancipated minors (15-17 years of age) with eligible children

Inclusion Criteria for eligible children:

* Biological children (of an index parent/caregiver) 18 months - 14 years of age with an unknown HIV status
* Non-biological children living in the same household as the index parent/caregivers where the child has a history of HIV exposure (where the mother is HIV-positive, of unknown status, unavailable for testing, or who is deceased)
* Biological children (of an index parent/caregiver) 18 months - 14 years of age, as well as non-biological children living in the same household as the index parent/caregiver where the child has a history of HIV exposure (where the mother is HIV-positive, of unknown status, unavailable for testing, or who is deceased), with a known previous HIV-negative status completed less than three months following the cessation of breastfeeding and whose parent/caregiver states that there is reason to suspect a new exposure

Inclusion criteria for participation in survey after completion of care giver-assisted oral fluid-based HIV screening:

• Adult index parents who complete the oral-based HIV screening with at least one eligible child, regardless of screening result.

Exclusion Criteria for Index parent/caregivers:

* Adults answering "yes" to any of the first three intimate partner violence (IPV) risk assessment questions
* Adults answering "yes", "maybe" or I don't know" to the fourth IPV question
* Those unable to provide independent informed consent due to mental disability or other limitations (as deemed by study staff)

Exclusion Criteria for eligible children:

* Children <18 months of age
* Children 18 months - 14 years of age with a known HIV-positive status
* Biological children (of an index parent/caregiver) 18 months - 14 years of age where the child has a history of HIV exposure (where the mother is HIV-positive, of unknown status, unavailable for testing, or who is deceased), with previous known HIV-negative status completed less than three months following the cessation of breastfeeding and whose parent/caregiver states that they have no reason to suspect a new exposure
* Non-biological children living in the same household as the index parent/caregiver age where the child has a history of HIV exposure (where the mother is HIV-positive, of unknown status, unavailable for testing, or who is deceased), with previous known HIV-negative status completed less than three months following the cessation of breastfeeding and whose parent/caregiver states that they have no reason to suspect a new exposure
* Children still breastfeeding
* Children with cessation of breastfeeding < 3 months

Exclusion criteria for participation in survey after completion of oral-based HIV screening:

• Adult index parent/caregivers who do not complete the oral-based HIV screening with at least one eligible child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At the 32 PEPFAR-supported government health facilities, eligible adult index parents and their eligible children will be recruited during post-test counseling sessions when they are newly-diagnosed as HIV-positive, and/or at the ART clinic and/or mother-baby care point (MBCP).
Sampling Method: Non-Probability Sample
Enrollment: 4865 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Estimate the acceptability of implementing caregiver-assisted oral fluid-based HIV screening of children as part of index testing services for HIV-positive adults. | 6 months
  * Proportion of eligible index parent/caregivers (disaggregated by sex) that accepted an oral fluid-based HIV screening kit as part of innovative index testing services for their eligible children when first offered.
  * Proportion of eligible index parent/caregivers (disaggregated by sex) that accepted an oral fluid-based HIV screening kit as part of innovative index testing services for their eligible children when they returned for a subsequent visit.
  * Proportion of eligible children (i.e. unknown HIV status) screened with an oral fluid-based HIV screening kit.
Estimate the feasibility of implementing caregiver-assisted oral fluid-based HIV screening for children as part of index testing services for HIV-positive adults. | 6 months
  * Proportion of index parent/caregivers who reported that the caregiver-assisted oral fluid-based HIV screening kit to screen children for HIV was easy to use.
  * Proportion of index parent/caregivers who reported needing additional assistance with administering the oral fluid-based HIV screening kit.
  * Proportion of index parent/caregivers who reported adverse events related to the use of caregiver-assisted oral fluid-based HIV screening kits to screen their children for HIV.
Estimate the effectiveness of caregiver-assisted oral fluid-based HIV screening on testing yield, return to clinic, and linkage to ART for newly identified CLHIV. | 6 months
  * Proportion of eligible children screened reactive through a caregiver-assisted oral fluid-based HIV screening kit (i.e., yield).
  * Proportion of eligible children who screened reactive through a caregiver-assisted oral fluid-based HIV screening kit who received confirmatory testing, within 1 day, 1 week, 1 month of their reactive screen.
  * Proportion of eligible children who screened reactive through a caregiver-assisted oral fluid-based HIV screening kit who were started on ART within 1 day, 1 week, 1 month of their confirmatory test.
  * Proportion of index parent/caregivers who were offered an oral fluid-based test kit to screen their eligible children for HIV used it.

SECONDARY OUTCOMES:
Estimate the cost of caregiver-assisted oral fluid-based HIV screening compared to the standard cost of the existing referral to testing program, from the perspective of the health care provider. | 6 months
  Comparative costs between oral fluid-based screening and the costs of the existing referral to testing program, from the perspective of the health care provider.

CONTACTS AND LOCATIONS:
Overall Officials: Carl C Stecker, EdD, Principal Investigator — Catholic Relief Services - USCCB
Locations (32):
- Uganda (32):
  - Bugiri Hospital, Bugiri, Bugiri District
  - Nankoma HC IV, Bugiri, Bugiri District
  - Kabuyanda HC IV, Kabuyanda, Isingiro District
  - Rwekubo HC IV, Kahirimbi, Isingiro District
  - Buremba HC III, Kazo, Kazo District
  - Kazo HC IV, Kazo, Kazo District
  - Butunduzi HC III, Kyenjojo, Kyenjojo District
  - Kigarale HC III, Kyenjojo, Kyenjojo District
  - Kasaali HC III, Kyotera, Kyotera District
  - Barr HC III, Lira, Lira District
  - Lira Regional Ref Hospital, Lira, Lira District
  - Luwero HC IV, Kampala, Luwero District
  - St. Luke Namaliga HC III, Kampala, Luwero District
  - Kinoni HC III, Bukoto, Lwengo District
  - Kiwangala HC III, Mbirizi, Lwengo District
  - Kiyumba HC IV, Bukoto, Masaka District
  - Buwunga HC III, Masaka, Masaka District
  - Mbarara Regional Ref Hospital, Mbarara, Mbarara District
  - Nyamityobora HC II, Mbarara, Mbarara District
  - Kyantungo HC IV, Mityana, Mityana District
  - Mityana Hospital, Mityana, Mityana District
  - Mubende Kasambya HC III, Mubende, Mubende District
  - Nabingoola HC III, Nabingora, Mubende District
  - Mukono Cou HC IV, Mukono, Mukono District
  - Seeta-Nazigo HC III, Nakisunga, Mukono District
  - Kitwe HC IV, Kitwe, Ntungamo District
  - Ntungamo HC IV, Ntungamo, Ntungamo District
  - Lwamaggwa HC III, Rakai, Rakai District
  - Rakai Hospital, Rakai, Rakai Distsrict
  - Kajjansi HC III, Busiro, Wakiso District
  - Kasangati HC IV, Kasangati, Wakiso District
  - Mitukula HC III, Kyotera

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gross J, Tumwesigye NM, Mutembo S, Moyo N, Mukose A, Chilyabanyama O, Matoba J, Parris K, Lee B, Churchill T, Williamson D, Pals S, Biribawa C, Kagaayi J, Ndubani P, Okello F, Zyambo Z, Taasi G, Magongo EN, Munthali G, Mwiya M, Nazziwa E, Awor AC, Itoh M, Boyd AM, Macleod D, Rivadeneira E, Oliver D, Ferrand RA, Stecker C; FASTER Study Team. Acceptability, feasibility, and effectiveness of caregiver-assisted HIV self-testing among children using an oral mucosal test in Uganda and Zambia: a prospective interventional study. Lancet HIV. 2025 May;12(5):e325-e337. doi: 10.1016/S2352-3018(25)00005-0. PMID 40316402